CLINICAL TRIAL: NCT01483898
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study To Evaluate The Efficacy, Safety, And Tolerability Of Ixmyelocel-T In Subjects With Critical Limb Ischemia And No Options For Revascularization
Brief Title: An Efficacy and Safety Study of Ixmyelocel-T in Patients With Critical Limb Ischemia (CLI)
Acronym: REVIVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vericel Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABI 55-1009-1
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Critical Limb Ischemia
Keywords: critical limb ischemia; REVIVE; peripheral vascular disease; CLI; PAD; MSC; stem cells; cell therapy
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ixmyelocel-T (Experimental)
  Interventions: Biological: Ixmyelocel-T
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Ixmyelocel-T — On Day 14, 20 intramuscular injections of ixmyelocel-T on pre-identified index leg.
  Arms: ixmyelocel-T
Other: Placebo — On Day 14, 20 intramuscular injections of vehicle control on pre-identified index leg.
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the efficacy and safety of ixmyelocel-T, a patient-specific expanded multicellular therapy, for the treatment of patients with critical limb ischemia (CLI). The study is a randomized, vehicle controlled (placebo)study in CLI patients who have no option for revascularization procedures. All patients randomized will undergo a small volume bone marrow aspiration in a 15-minute outpatient or in-office procedure. All patients will receive injections of either ixmyelocel-T or vehicle-control into their pre-identified index leg. Patients will be followed for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Males and nonpregnant, nonlactating females
* Ages 35 to 90 years of age
* Diagnosis of CLI with tissue loss (corresponding to Rutherford Category 5; see Appendix B) having an ulcer size of at least 0.5 cm2, a smaller sized ulcer penetrating into the subcutaneous tissue, and/or gangrene (dry). In addition, the subject must have ONE of the following documented at screening:

  * Ankle systolic pressure < 70 mm Hg
  * Toe systolic pressure < 50 mm Hg
  * TcPO2 < 30 mm Hg (in a supine position)
* Subjects must have no reasonable standard-of-care options for surgical or endovascular revascularization interventions
* Subjects must have the following:

  * A narrative documenting the reasons why the site vascular specialist considers the subject "no option". A vascular specialist will be the principal investigator (PI) or subinvestigator and is defined as: vascular surgeon, interventional cardiologist, certified vascular medicine specialist, or interventional radiologist; AND
  * Secondary confirmation by an independent Eligibility Review Committee (ERC; see Section 8.1) after review of appropriate documents including, but not limited to: imaging results, medical records, surgical history, site vascular specialist narrative documenting reasons for "no option," and/or lab reports.
* Major amputation in the index leg or death is not anticipated within 3 months of screening in the opinion of the vascular specialist (who must be the PI or subinvestigator)
* In the opinion of the investigator, the subject is controlled on medical therapy indicated for CLI (unless there is a documented contraindication or intolerance)
* Subject is current with all age-appropriate American Cancer Society (ACS) or similar (e.g., United States Preventative Service Task Force) screening guidelines
* Given medical history and concurrent medication, the subject is an acceptable candidate for bone marrow aspiration and intramuscular injection procedures in the opinion of the Investigator
* Subject is willing and able to comply with the scheduled visits, aspiration/injection procedure, wound care instructions treatment plan, and other study procedures for the duration of the study
* Provide a personally-signed and dated informed consent document indicating that the subject (or a legally-acceptable representative, if permitted by the site's Investigational Review Board [IRB]) has been informed of all pertinent aspects of the study

Exclusion Criteria:

Patients presenting with any of the following will not be randomized:

Disease-specific:

* Failed open surgical revascularization (on index leg) within 4 weeks of screening Visit 1
* Acute limb-threatening ischemia, trauma, known non-atherosclerotic vascular disease (e.g., temporal/giant cell arteritis, Takayasu's arteritis, Raynaud's occlusive disease, Buerger's disease), embolic disease, aortoiliac disease with > 50% stenosis, or history of hypercoagulable states
* Advanced CLI (i.e., nonsalvageable) defined as Rutherford Category 6
* Clinical evidence of invasive infection in index leg (e.g., cellulitis, osteomyelitis, wet gangrene)
* At screening, non-heel wound size of > 20 cm2 (excluding toe gangrene); or wounds on the heel > 10 cm2 on the index leg as measured by the Wound Core Lab (WCL) from photographs (and/or acetates) provided by the site
* Previous amputation at or above the talus in the index leg Medical History
* Hemoglobin A1c (HbA1c) ≥ 10% at screening
* Diabetic subjects with uncontrolled or untreated proliferative retinopathy as determined by dilated eye exam (by qualified eye care professional as per American Diabetes Association guidelines)
* Blood clotting disorder not caused by medication (e.g., thrombophilia)
* Active non-basal cell cutaneous malignancy requiring surgery, chemotherapy, and/or radiation in the past 12 months
* Current documented drug or alcohol abuse that would interfere with the subject's compliance with study procedures
* Known allergies to any equine, porcine, or bovine products
* Body mass index (BMI) ≥ 50 kg/m2 at screening
* Established chronic kidney disease (CKD) requiring dialysis (Stage 5); estimated creatinine clearance < 15 mg/mL/min at screening
* Systolic blood pressure (SBP) > 200 mm Hg or diastolic blood pressure (DBP) > 120 mm Hg or papilledema noted via ophthalmoscope at screening physical exam
* Within 3 months prior to screening, a clinically significant history of cardiac disease

Laboratory Parameters:

* Abnormal laboratory values (performed at central lab) at screening:

  * Platelets < 50,000 μL
  * Aspartate aminotransferase/alanine aminotransferase (AST/ALT) > 3 times the upper limit of normal (ULN)
  * Human immunodeficiency virus 1 (HIV 1), HIV 2, or syphilis positive (rapid plasma reagin [RPR])
  * Active hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV); Exclusionary Procedures, Devices, or Medication
* Exposure to immunosuppressive therapy for oncologic or chronic non-oncologic reasons in the prior 12 months or expected requirement over the course of the study (e.g., chemotherapy, radiation therapy, methotrexate)
* Concurrent participation in another clinical trial or receiving experimental medication within 30 days of screening or having previously been exposed to Aastrom's ixmyelocel T product [previously known as tissue repair cells (TRC), cardiac repair cells (CRC), vascular repair cells (VRC)]
* On the index leg, use of concomitant wound treatments not currently approved for ischemic wound-healing within 30 days prior to screening or plans to initiate new, nonstandard-of-care treatments to the index leg during the study

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-02; Primary Completion 2014-03-25 (Actual); Study Completion 2014-03-25 (Actual)

PRIMARY OUTCOMES:
Amputation free survival (AFS) at 12 months post-injection | 12 months
  The primary objective will be to assess the efficacy of ixmyelocel-T compared to placebo (vehicle control) on AFS at 12 months post-injection in CLI patients with no options for revascularization. Amputation free survival is defined as time to the first occurrence of either major amputation (above the talus) in the index leg or all-cause mortality (death).

SECONDARY OUTCOMES:
Percent of patients with adverse events | 18 months
  A secondary objective will be to evaluate the overall safety and tolerability of ixmyelocel-T versus placebo in patients with CLI from time of aspiration through 18 months post-treatment/follow-up by % of patients with adverse events.
Percent of patients with complete wound closure by Month 12 | 12 months
  A secondary objective is to assess the percent of patients with at least 1 ischemic wound on the index leg that is present at Visit 3 (preinjection) having complete closure by Month 12.
Percent of patients experiencing a major cardiac event (MACE) by Months 6, 12, and 18 | 6, 12 and 18 months
  % of patients experiencing a MACE event defined as cardiovascular mortality, myocardial infarction, chest pain requiring hospitalization, or stroke.

CONTACTS AND LOCATIONS:
Locations (86):
- United States (86):
  - Cardiology PC, Birmingham, Alabama
  - Cardio-Thoracic Surgeons, P.C., Birmingham, Alabama
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Arizona Heart Institute, Phoenix, Arizona
  - Carl T. Hayden VA Medical Center, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Arkansas Primary Care Clinic, P.A., Little Rock, Arkansas
  - Central Arkansas Veteran's Healthcare System, Little Rock, Arkansas
  - John Muir Medical Center - Concord Campus, Concord, California
  - VA Loma Linda Healthcare, Loma Linda, California
  - UCLA Gonda Venous Center & Ambulatory Procedure Unit, Los Angeles, California
  - Sutter Medical Group - Cardiology, Sacramento, California
  - University of California San Diego Medical Center, San Diego, California
  - Kaiser Permanente Medical Center, San Diego, California
  - University of California San Francisco - Division of Vascular and Endovascular Surgery, San Francisco, California
  - University of Colorado Denver - Anschutz Medical Campus, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Bethesda Memorial Hospital - Clinical Research Center, Boynton Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Florida Research Network, LLC, Gainesville, Florida
  - Malcom Randall Veterans Affairs Medical Center, Gainesville, Florida
  - First Coast Cardiovascular Institute, P.A., Jacksonville, Florida
  - University of Miami Hospital, Miami, Florida
  - Orlando Health, Orlando, Florida
  - Baptist Hospital, Pensacola, Florida
  - Cardiology Consultants, Pensacola, Florida
  - Grove Place Surgery Center, Vero Beach, Florida
  - Vascular Surgical Associates, P.C., Marietta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago - Clinical Sciences North, Chicago, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Indiana/Ohio Heart, Fort Wayne, Indiana
  - St. Vincent Medical Group, Inc., Indianapolis, Indiana
  - Heartland Vascular Medicine and Surgery, Windsor Heights, Iowa
  - Ochsner Clinic foundation, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Union Memorial Hospital, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - UMASS Memorial Health Care, Worcester, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - Cardiology and Vascular Associates, P.C., Berkley, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - John D. Dingell VA Medical Center, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan Vascular Research Center, Flint, Michigan
  - Integrated Vascular Vein Center of Michigan, Grand Blanc, Michigan
  - Michigan CardioVascular Institutue at Covenant Medical Center, Saginaw, Michigan
  - Saint Joseph Mercy Hospital, Ypsilanti, Michigan
  - Abbott Northwestern Hospital / Minneapolis Heart Institute-Vascular Clinic, Minneapolis, Minnesota
  - Minneapolis VA Health Care System, Minneapolis, Minnesota
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Hattiesburg Clinic, P.A., Hattiesburg, Mississippi
  - Saint Luke's Hospital, Kansas City, Missouri
  - Omaha VAMC, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Vascular Access Center of West Orange, West Orange, New Jersey
  - University of Buffalo Surgeons Inc., Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Jobst Vascular Institute, Toledo, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Veterans' Administration Medical Center, Pittsburgh, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - DFW Vascular Group, LLP, Dallas, Texas
  - Texas Heart Institute at St. Luke's Episcopal Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - Audie L Murphy VA Hospital - Pathology Laboratory, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - Swedish Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Cascade Vascular Associates, P.S., Tacoma, Washington
  - Charleston Area Medical Center - Memorial Hospital, Charleston, West Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Columbia Saint Mary's, Milwaukee, Wisconsin
  - Wheaton Franciscan Medical Group, Inc., Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Aastrom Biosciences Homepage — http://www.aastrom.com/
- See also: Vascular web provided by The Society for Vascular Surgery — http://www.vascularweb.org
- See also: Legs For Life — http://www.legsforlife.org
- See also: University of California, Davis — http://www.ucdmc.ucdavis.edu/vascular/diseases/cli.html
- See also: Mayo Clinic — http://www.mayoclinic.com/health/peripheral-arterial-disease/DS00537